CLINICAL TRIAL: NCT01028508
Title: Prolonging Remission in Depressed Elderly (PRIDE)
Acronym: PRIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 09-0429; U01MH055495 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Depression; ECT; electroconvulsive therapy; mood disorders; continuation ECT; continuation pharmacotherapy; geriatric; elderly; lithium; venlafaxine
MeSH Terms: conditions — Depression; Mood Disorders | interventions — Lithium; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHARM (Active Comparator): lithium and venlafaxine
  Interventions: Drug: lithium and Venlafaxine
- STABLE (Experimental): ECT + VLF + Li
  Interventions: Procedure: ECT

INTERVENTIONS:
Drug: lithium and Venlafaxine — Drug: VLF Target dose 225 mg/day Drug: Li Target serum concentration 0.7 mEq/l
  Arms: PHARM
Procedure: ECT — Procedure: ECT RUL ultra brief pulse ECT, 4 treatments in one month and then treatment on an as-needed basis for 5 months Drug: VLF Target dose 225 mg/day Drug: Li Target serum concentration 0.7 mEq/l
  Arms: STABLE

SUMMARY:
This study will determine whether medications alone or medications and electroconvulsive therapy (ECT) work best to prevent depressive relapse and to improve quality of life for older people with severe mood disorders.

DETAILED DESCRIPTION:
While advances have been made in the acute treatment of geriatric depression, failure to maintain remission following successful treatment remains a major public health problem. In particular, loss of antidepressant response can result in ongoing functional impairment and increased risk of suicide. This is especially salient for severe and/or treatment resistant illness, even after successful ECT.

This trial builds upon the work of the Consortium for Research in Electroconvulsive Therapy (CORE) group that showed that continuation ECT and combination pharmacotherapy were equally effective in preventing relapse following response to acute ECT. We are now testing whether combined pharmacotherapy and ECT, individualized according to patient response, will be more effective in maintaining remission in depressed older adults than pharmacotherapy alone. Moving beyond the traditional fixed schedule for continuation ECT, we are introducing a novel Symptom-Titrated Algorithm-Based Longitudinal ECT (STABLE) regimen. The STABLE algorithm ensures that the timing of ECT treatments is based upon clinical need, helping to achieve the dual goals of adequately treating people showing early signs of symptom re-emergence, while preventing the over-treatment of patients who may be in a stable remission. The continuation therapy "usual care" comparator arm is the combination pharmacotherapy of Li plus VLF (PHARM).

At 7 sites, 322 patients will receive an acute course of right unilateral (RUL) ECT augmented by standardized medication (Phase I); 188 remitters are randomly assigned to one of the 2 groups and followed for 6 months (Phase II). To balance the amount of clinical contact, the schedule of clinic and telephone ratings will be identical for patients in both the PHARM and STABLE arms. For both groups, relapse is defined as Hamilton Rating Scale for Depression-24 (HRSD24) scores >21 at two consecutive time points, suicidality, or psychiatric hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depressive episode, unipolar, based on the Mini-International Neuropsychiatric Interview (M.I.N.I) for DSM-IV
* ECT is clinically indicated

Exclusion Criteria:

* Lifetime history of bipolar affective disorder, schizophrenia, schizoaffective disorder, or mental retardation
* Current diagnosis of delirium, dementia, or substance abuse/dependence in past 6 months as defined by DSM-IV-TR criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2010-01; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at every week
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 2
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 4
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 5
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 6
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 7
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 8
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 9
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 10
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 11
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 12
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 13
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 14
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 15
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 16
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 17
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 18
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 19
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 20
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 21
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 22
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured by a telephone interview at week 23
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23
Long-term antidepressant efficacy (Hamilton Rating Scale for Depression) | Measured at clinic visits at week 24
  Long-term antidepressant efficacy (Hamilton Rating Scale for Depression)
  Measured at clinic visits at baseline and weeks 2, 4, 6, 8, 10,12,14,16, 18, 20, 22, 24.
  Measured by a telephone interview at weeks 5, 7, 9, 11, 13, 15, 17, 19, 21, 23

SECONDARY OUTCOMES:
Level of functioning (SF-36) | Measured at baseline
  Level of functioning (SF-36) measured at baseline and weeks 4, 8, 12, 16, 20, 24
Level of functioning (SF-36) | Measured at week 4
  Level of functioning (SF-36) measured at baseline and weeks 4, 8, 12, 16, 20, 24
Level of functioning (SF-36) | Measured at week 8
  Level of functioning (SF-36) measured at baseline and weeks 4, 8, 12, 16, 20, 24
Level of functioning (SF-36) | Measured at week 12
  Level of functioning (SF-36) measured at baseline and weeks 4, 8, 12, 16, 20, 24
Level of functioning (SF-36) | Measured at week 16
  Level of functioning (SF-36) measured at baseline and weeks 4, 8, 12, 16, 20, 24
Level of functioning (SF-36) | Measured at week 20
  Level of functioning (SF-36) measured at baseline and weeks 4, 8, 12, 16, 20, 24
Level of functioning (SF-36) | Measured at week 24
  Level of functioning (SF-36) measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at baseline
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 2
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 4
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 8
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 10
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 12
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 14
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 16
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 18
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 20
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 22
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (Mini Mental State Examination [MMSE]) | Measured at week 24
  Tolerability (Mini Mental State Examination [MMSE]) Measured at baseline, and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) | Measured at baseline
  Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) Measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) | Measured at week 4
  Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) Measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) | Measured at week 8
  Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) Measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) | Measured at week 12
  Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) Measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) | Measured at week 16
  Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) Measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) | Measured at week 20
  Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) Measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) | Measured at week 24
  Tolerability (California Verbal Learning Test [CVLT-II], Autobiographical Memory Interview-Short Form [AMI-SF]) Measured at baseline and weeks 4, 8, 12, 16, 20, 24
Tolerability (Trail Making Tests, DRS-IP and Delis-Kaplan Executive Function System, Verbal Fluency | Measured at baseline
  Tolerability (Trail Making Tests, DRS-IP and Delis-Kaplan Executive Function System, Verbal Fluency Measured at baseline and weeks 12, 24
Tolerability (Trail Making Tests, DRS-IP and Delis-Kaplan Executive Function System, Verbal Fluency | Measured at weeks 12
  Tolerability (Trail Making Tests, DRS-IP and Delis-Kaplan Executive Function System, Verbal Fluency Measured at baseline and weeks 12, 24
Tolerability (Trail Making Tests, DRS-IP and Delis-Kaplan Executive Function System, Verbal Fluency | Measured at weeks 24
  Tolerability (Trail Making Tests, DRS-IP and Delis-Kaplan Executive Function System, Verbal Fluency Measured at baseline and weeks 12, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at baseline
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 2
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 4
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 6
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 8
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 10
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 12
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 14
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 16
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 18
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 20
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 22
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) | Measured at week 24
  Safety (Udvalg for Kliniske Undersogelser [UKU] Side Effects Rating Scale) Measured at baseline and weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kellner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (10):
- United States (10):
  - Georgia Regents University, Augusta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Hoboken University Medical Center (MSSM satellite site), Hoboken, New Jersey
  - The Zucker Hillside Hospital North Shore-LIJ Health System, Glen Oaks, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University/New York State Psychiatric Institute, New York, New York
  - Weill Cornell Medical College, White Plains, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Medical Center, Winston-Salem, North Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Background] Kellner CH, Knapp RG, Petrides G, Rummans TA, Husain MM, Rasmussen K, Mueller M, Bernstein HJ, O'Connor K, Smith G, Biggs M, Bailine SH, Malur C, Yim E, McClintock S, Sampson S, Fink M. Continuation electroconvulsive therapy vs pharmacotherapy for relapse prevention in major depression: a multisite study from the Consortium for Research in Electroconvulsive Therapy (CORE). Arch Gen Psychiatry. 2006 Dec;63(12):1337-44. doi: 10.1001/archpsyc.63.12.1337. PMID 17146008
- [Background] Sackeim HA, Haskett RF, Mulsant BH, Thase ME, Mann JJ, Pettinati HM, Greenberg RM, Crowe RR, Cooper TB, Prudic J. Continuation pharmacotherapy in the prevention of relapse following electroconvulsive therapy: a randomized controlled trial. JAMA. 2001 Mar 14;285(10):1299-307. doi: 10.1001/jama.285.10.1299. PMID 11255384
- [Derived] Lisanby SH, McClintock SM, McCall WV, Knapp RG, Cullum CM, Mueller M, Deng ZD, Teklehaimanot AA, Rudorfer MV, Bernhardt E, Alexopoulos G, Bailine SH, Briggs MC, Geduldig ET, Greenberg RM, Husain MM, Kaliora S, Latoussakis V, Liebman LS, Petrides G, Prudic J, Rosenquist PB, Sampson S, Tobias KG, Weiner RD, Young RC, Kellner CH; Prolonging Remission in Depressed Elderly (PRIDE) Work Group. Longitudinal Neurocognitive Effects of Combined Electroconvulsive Therapy (ECT) and Pharmacotherapy in Major Depressive Disorder in Older Adults: Phase 2 of the PRIDE Study. Am J Geriatr Psychiatry. 2022 Jan;30(1):15-28. doi: 10.1016/j.jagp.2021.04.006. Epub 2021 May 17. PMID 34074611
- [Derived] Lisanby SH, McClintock SM, Alexopoulos G, Bailine SH, Bernhardt E, Briggs MC, Cullum CM, Deng ZD, Dooley M, Geduldig ET, Greenberg RM, Husain MM, Kaliora S, Knapp RG, Latoussakis V, Liebman LS, McCall WV, Mueller M, Petrides G, Prudic J, Rosenquist PB, Rudorfer MV, Sampson S, Teklehaimanot AA, Tobias KG, Weiner RD, Young RC, Kellner CH; CORE/PRIDE Work Group. Neurocognitive Effects of Combined Electroconvulsive Therapy (ECT) and Venlafaxine in Geriatric Depression: Phase 1 of the PRIDE Study. Am J Geriatr Psychiatry. 2020 Mar;28(3):304-316. doi: 10.1016/j.jagp.2019.10.003. Epub 2019 Oct 12. PMID 31706638
- [Derived] McCall WV, Lisanby SH, Rosenquist PB, Dooley M, Husain MM, Knapp RG, Petrides G, Rudorfer MV, Young RC, McClintock SM, Mueller M, Prudic J, Greenberg RM, Weiner RD, Bailine SH, Youssef NA, McCloud L, Kellner CH; CORE/PRIDE Work Group. Effects of continuation electroconvulsive therapy on quality of life in elderly depressed patients: A randomized clinical trial. J Psychiatr Res. 2018 Feb;97:65-69. doi: 10.1016/j.jpsychires.2017.11.001. Epub 2017 Nov 16. PMID 29195125
- [Derived] McCall WV, Lisanby SH, Rosenquist PB, Dooley M, Husain MM, Knapp RG, Petrides G, Rudorfer MV, Young RC, McClintock SM, Mueller M, Prudic J, Greenberg RM, Weiner RD, Bailine SH, Riley MA, McCloud L, Kellner CH; CORE/PRIDE Work Group. Effects of a Course of Right Unilateral Ultrabrief Pulse Electroconvulsive Therapy Combined With Venlafaxine on Insomnia Symptoms in Elderly Depressed Patients. J Clin Psychiatry. 2018 Mar/Apr;79(2):16m11089. doi: 10.4088/JCP.16m11089. PMID 28742292
- [Derived] McCall WV, Lisanby SH, Rosenquist PB, Dooley M, Husain MM, Knapp RG, Petrides G, Rudorfer MV, Young RC, McClintock SM, Mueller M, Prudic J, Greenberg RM, Weiner RD, Bailine SH, Riley MA, McCloud L, Kellner CH; CORE/PRIDE Work Group. Effects of a right unilateral ultrabrief pulse electroconvulsive therapy course on health related quality of life in elderly depressed patients. J Affect Disord. 2017 Feb;209:39-45. doi: 10.1016/j.jad.2016.11.003. Epub 2016 Nov 11. PMID 27886569
- [Derived] Kellner CH, McClintock SM, McCall WV, Petrides G, Knapp RG, Weiner RD, Young RC, Greenberg RM, Rudorfer MV, Ahle GM, Liebman LS, Lisanby SH; CORE/PRIDE Group. Brief pulse and ultrabrief pulse right unilateral electroconvulsive therapy (ECT) for major depression: efficacy, effectiveness, and cognitive effects. J Clin Psychiatry. 2014 Jul;75(7):777. doi: 10.4088/JCP.14lr08997. No abstract available. PMID 25093475